CLINICAL TRIAL: NCT03163394
Title: HD5 Levels in Catheter Versus Bag Urine Specimens in Young Children for the Diagnosis of UTI
Status: Terminated | Type: Observational
Why Stopped: Did not enroll enough patients for study
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Kristy Morse, Principal Investigator, Le Bonheur Children's Hospital
Other Study IDs: HD52017
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urinary tract infections (UTIs) are a common cause of bacteremia and serious bacterial infections in young children (2-24 months of age). Because these children are usually unable to say what symptoms they are experiencing, UTIs are diagnosed through testing. Current testing of urine samples require a catheter or suprapubic aspiration performed for urine collection for infections markers to be reliable. Bag specimens often have varying results that can be poor in sensitivity and specificity depending on what component of the urine test one is looking at. Catheter and aspiration testing can be anxiety-provoking to parents, be painful for patients and even introduce bacteria into the bladder. An antimicrobial peptide called alpha human defensin-5 (HD5) is produced by the uroepithelium in response to infection. HD5 has been studied in the urine and does increase in actual UTIs. This study will look at children 1 to 24 months of age and again study levels of HD5 in culture positive UTIs versus urine negative for UTI. This study will also determine if collection method alters HD5 levels. We will measure HD5 levels in the urine from a bag specimen and a catheter specimen in the same patient.

Our primary objective is to determine the sensitivity and specificity of HD5 measured in urine collected by bag and catheter in the same patient for the diagnosis of UTI in children between the age 1 to 24 months presenting with febrile illness and suspected UTI.

DETAILED DESCRIPTION:
Pediatric urinary tract infections (UTIs) are a common diagnosis and account for greater than 500,000 emergency department (ED) visits each year in the US. Although prevalence varies by age, gender, ethnicity and circumcision status, the overall prevalence is cited between 5% to 13.8%. UTIs also account for a large number of pediatric hospital admissions with up to 50,000 children admitted per year, 40% of which occurring in children under the age of 1 year. In children under the age of two, diagnosis of UTI is difficult as patients are unable to verbalize complaints and often present with only fever or other nonspecific symptoms such as vomiting. UTIs are the leading cause of occult bacteremia and serious bacterial infection in the 2-24 month age range.

A definitive diagnosis of UTI is made when a patient has pyuria and/or bacteriuria with a positive urine culture. For non-toilet trained children who have urine collected by either suprapubic aspiration (SPA) or bladder catheterization, a urine culture is considered positive if a single uropathogenic organism of at least 50,000 colony forming units (CFU) per mL is recovered. Identification of a uropathogen by culture can take up to 48 hours to be completed which delays treatment and risks progression of infection if antibiotics are not given empirically. Commonly, clinicians use urine microscopy and dipstick for quick diagnosis to enable early empiric treatment of UTIs. However, the components of the urinalysis are limited in sensitivity and specificity even for specimens of high quality such as those obtained by catheterization or suprapubic tap. The main components of urine dipstick testing are leukocyte esterase (LE) and nitrite levels in urine. The LE test has a sensitivity of 94% when combined with clinical suspicion for UTI, but a specificity of only 83%. False positives for UTI occur when LE is positive in the child who has pyuria for other reasons besides infection, for example, in urethritis or Kawasaki disease. False negatives can occur in young children because the pattern of more frequent urination allows less time to mount an adequate inflammatory response to bacteria. Nitrites have a low sensitivity in young children (53%) due to frequent voiding not allowing sufficient time (up to 4 hours) for production of nitrites by bladder-dwelling bacteria; however, specificity is high (98%) making this a good test to rule in UTI. Sensitivity and specificity of urine microscopy for WBCs and bacteria are worse than for LE with pyuria (5 or more WBC/high power field on a spun sample or >10 WBC/hpf on an un-spun sample) having a sensitivity and specificity of 73% and 81% respectively. Presence of bacteria on microscopy has a sensitivity and specificity of 81% and 83% respectively. The resulting over- and under-treatment for false positive and negative urinalyses leads to increased costs, antibiotic resistance and unnecessary adverse events from antibiotics. The inaccuracy of the traditional urinalysis on bagged urine samples is much greater than for catheter specimens. These specimens suffer from false positives results for leukocyte esterase and cultures at rates up to 75-88% because of contamination by urogenital flora and white blood cells present on the perineum.

As a result of the poor performance characteristics of routine urinalyses on bag specimens, a sample obtained by catheterization in children who are not yet toilet-trained is required even for UTI screening. This is invasive and painful for the child, causes anxiety for the family, leads to urethral trauma and can even introduce bacteria into the urinary system. Recent research describes a new two-step technique of obtaining urine samples of screening for UTI on these young patients. First, a bagged urine sample is taken, and if suspicious for UTI by urinalysis, the patient then is catheterized for culture. One study showed that this technique decreased the number of catheterizations by 33%; however, given the low specificity of the urinalyses on bag specimens, there is still substantial room for reductions in unnecessary bladder catheterizations.

New urinary biomarkers hold promise to improve screening accuracy for UTIs. Watson et al. investigated antimicrobial peptides (AMPs) as urinary biomarkers of UTIs in children. One specific AMP, derived from the epithelium, is human alpha-defensin 5 (HD5). This AMP is produced by intestinal Paneth cells, the female genital tract and the uroepithelium. HD5 was found to have mean concentration significantly higher in the urine from culture-positive compared to culture-negative specimens. When used in combination with LE, HD5 increased the specificity of the LE-only test by 6% without decreasing the sensitivity (97% for LE > trace). This study determined the optimal cut-off value of 174 pg/mg creatinine to declare sample positive. Because HD5 is not derived from white blood cells, its presence is not affected by the presence or absence of WBCs in the urine to accurately identify urinary inflammation. While the authors of this study examined results from both clean-catch and catheterized specimens, they did not analyze samples collected by both techniques from the same patient.

Identification and validation of biomarkers with improved performance characteristics could reduce over-treatment of UTIs; validating such biomarkers on bag urine specimens has the further benefit of reducing the need for catheterization to provide urine to screen for UTI in a relatively unselected population of young children who have fever without a focus. We propose to compare the use of HD5 in bag versus catheter urine samples on children 1 to 24 months of age to determine if the biomarker has similarly high sensitivity and specificity to the original study in both specimen types. Eliminating the need for urine culture would also save on costs for children whose rapid testing does not suggest UTI. Reducing the number of catheterizations performed on young children will decrease the number of painful procedures, prevent introduction of bacteria in the urinary tract and decrease parental anxiety.

ELIGIBILITY:
Inclusion Criteria:

Patient is between 1 to 24 months of age Patient has reported or measured fever >38.5 degrees C (101.3 degrees F)

Exclusion Criteria:

RSV Positive at time of urine collection Flu Positive at time of urine collection Known GU abnormality Neurogenic bladder Frequent catheterizations Indwelling catheter Antibiotics in the last 7 days

Ages: 1 Month to 24 Months | Sex: All
Age Groups: Child
Study Population: Children between the age of 1 to 24 months that present to the LeBonheur Emergency Room with fever of 38.5 degrees Celsius by report or on measurement will have urine bag placed. If patient has urinalysis and urine culture ordered because of suspicion for UTI and patient has voided in the bag, then patient's family will be approached for research
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of HD5 as marker for UTI | 1 year
  The sensitivity and specificity of HD5 in determining urinary tract infections in bag versus catheter specimens in children aged 1 to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristy Morse, Principal Investigator — UTHSC
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Spencer JD, Schwaderer A, McHugh K, Hains DS. Pediatric urinary tract infections: an analysis of hospitalizations, charges, and costs in the USA. Pediatr Nephrol. 2010 Dec;25(12):2469-75. doi: 10.1007/s00467-010-1625-8. Epub 2010 Aug 14. PMID 20711740
- [Background] Subcommittee on Urinary Tract Infection, Steering Committee on Quality Improvement and Management; Roberts KB. Urinary tract infection: clinical practice guideline for the diagnosis and management of the initial UTI in febrile infants and children 2 to 24 months. Pediatrics. 2011 Sep;128(3):595-610. doi: 10.1542/peds.2011-1330. Epub 2011 Aug 28. PMID 21873693
- [Background] Sahsi RS, Carpenter CR. Evidence-based emergency medicine/rational clinical examination abstract. Does this child have a urinary tract infection? Ann Emerg Med. 2009 May;53(5):680-4. doi: 10.1016/j.annemergmed.2008.05.031. Epub 2008 Jul 21. No abstract available. PMID 19380042
- [Background] Williams GJ, Macaskill P, Chan SF, Turner RM, Hodson E, Craig JC. Absolute and relative accuracy of rapid urine tests for urinary tract infection in children: a meta-analysis. Lancet Infect Dis. 2010 Apr;10(4):240-50. doi: 10.1016/S1473-3099(10)70031-1. PMID 20334847
- [Background] Gorelick MH, Shaw KN. Screening tests for urinary tract infection in children: A meta-analysis. Pediatrics. 1999 Nov;104(5):e54. doi: 10.1542/peds.104.5.e54. PMID 10545580
- [Background] Lee HE, Kim DK, Kang HK, Park K. The diagnosis of febrile urinary tract infection in children may be facilitated by urinary biomarkers. Pediatr Nephrol. 2015 Jan;30(1):123-30. doi: 10.1007/s00467-014-2905-5. Epub 2014 Aug 16. PMID 25127917
- [Background] Glissmeyer EW, Korgenski EK, Wilkes J, Schunk JE, Sheng X, Blaschke AJ, Byington CL. Dipstick screening for urinary tract infection in febrile infants. Pediatrics. 2014 May;133(5):e1121-7. doi: 10.1542/peds.2013-3291. PMID 24777232
- [Background] Downs SM. Technical report: urinary tract infections in febrile infants and young children. The Urinary Tract Subcommittee of the American Academy of Pediatrics Committee on Quality Improvement. Pediatrics. 1999 Apr;103(4):e54. doi: 10.1542/peds.103.4.e54. PMID 10103346
- [Background] Schroeder AR, Chang PW, Shen MW, Biondi EA, Greenhow TL. Diagnostic accuracy of the urinalysis for urinary tract infection in infants <3 months of age. Pediatrics. 2015 Jun;135(6):965-71. doi: 10.1542/peds.2015-0012. PMID 26009628
- [Background] Schmidt B, Copp HL. Work-up of Pediatric Urinary Tract Infection. Urol Clin North Am. 2015 Nov;42(4):519-26. doi: 10.1016/j.ucl.2015.05.011. Epub 2015 Aug 4. PMID 26475948
- [Background] Bonadio WA. Urine culturing technique in febrile infants. Pediatr Emerg Care. 1987 Jun;3(2):75-8. doi: 10.1097/00006565-198706000-00003. PMID 3615238
- [Background] Kazi BA, Buffone GJ, Revell PA, Chandramohan L, Dowlin MD, Cruz AT. Performance characteristics of urinalyses for the diagnosis of pediatric urinary tract infection. Am J Emerg Med. 2013 Sep;31(9):1405-7. doi: 10.1016/j.ajem.2013.06.037. Epub 2013 Jul 26. PMID 23891600
- [Background] Whiting P, Westwood M, Watt I, Cooper J, Kleijnen J. Rapid tests and urine sampling techniques for the diagnosis of urinary tract infection (UTI) in children under five years: a systematic review. BMC Pediatr. 2005 Apr 5;5(1):4. doi: 10.1186/1471-2431-5-4. PMID 15811182
- [Background] Hay AD, Sterne JA, Hood K, Little P, Delaney B, Hollingworth W, Wootton M, Howe R, MacGowan A, Lawton M, Busby J, Pickles T, Birnie K, O'Brien K, Waldron CA, Dudley J, Van Der Voort J, Downing H, Thomas-Jones E, Harman K, Lisles C, Rumsby K, Durbaba S, Whiting P, Butler CC. Improving the Diagnosis and Treatment of Urinary Tract Infection in Young Children in Primary Care: Results from the DUTY Prospective Diagnostic Cohort Study. Ann Fam Med. 2016 Jul;14(4):325-36. doi: 10.1370/afm.1954. PMID 27401420
- [Background] Lavelle JM, Blackstone MM, Funari MK, Roper C, Lopez P, Schast A, Taylor AM, Voorhis CB, Henien M, Shaw KN. Two-Step Process for ED UTI Screening in Febrile Young Children: Reducing Catheterization Rates. Pediatrics. 2016 Jul;138(1):e20153023. doi: 10.1542/peds.2015-3023. Epub 2016 Jun 2. PMID 27255151
- [Background] Watson JR, Hains DS, Cohen DM, Spencer JD, Kline JM, Yin H, Schwaderer AL. Evaluation of novel urinary tract infection biomarkers in children. Pediatr Res. 2016 Jun;79(6):934-9. doi: 10.1038/pr.2016.33. Epub 2016 Feb 17. PMID 26885759
- [Background] Spencer JD, Hains DS, Porter E, Bevins CL, DiRosario J, Becknell B, Wang H, Schwaderer AL. Human alpha defensin 5 expression in the human kidney and urinary tract. PLoS One. 2012;7(2):e31712. doi: 10.1371/journal.pone.0031712. Epub 2012 Feb 16. PMID 22359618
- [Background] Spencer JD, Schwaderer AL, Becknell B, Watson J, Hains DS. The innate immune response during urinary tract infection and pyelonephritis. Pediatr Nephrol. 2014 Jul;29(7):1139-49. doi: 10.1007/s00467-013-2513-9. Epub 2013 Jun 5. PMID 23732397
- [Background] Caterino JM, Hains DS, Camargo CA, Quraishi SA, Saxena V, Schwaderer AL. A Prospective, Observational Pilot Study of the Use of Urinary Antimicrobial Peptides in Diagnosing Emergency Department Patients With Positive Urine Cultures. Acad Emerg Med. 2015 Oct;22(10):1226-30. doi: 10.1111/acem.12770. Epub 2015 Sep 16. PMID 26375724